CLINICAL TRIAL: NCT07093125
Title: An Observational Study on Rehabilitation Practices in the ICU for Critically Ill Patients Undergoing Invasive Mechanical Ventilation - Report (REPOrt)
Brief Title: Rehabilitation Practices in Critically Ill Patients Receiving Invasive Mechanical Ventilation in the Intensive Care Unit.
Acronym: REPOrt
Status: Not yet recruiting | Type: Observational
Sponsor: Universita degli Studi di Genova (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Denise Battaglini, Professor, Universita degli Studi di Genova
Other Study IDs: Liguria: 419/2024 - id 14164
Record Dates: First submitted 2025-05-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Pulmonary Rehabilitation; Intensive Care Units (ICUs); Quality of Life (QOL); Outcome Assessment; Extubation Failure; Mortality; Critical Care
Keywords: Pulmonary rehabilitation; Mechanical Ventilation; Intensive Care Unit (ICU); Rehabilitation Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients admitted in ICU and on mechanical ventilation for at least 48 hours: Adult patients who can be candidated to rehabilitation during ICU stay

SUMMARY:
This international, multicenter, observational study aims to describe rehabilitation practices in Intensive Care Units (ICUs) worldwide.

The primary objective is to provide an overview of current rehabilitation strategies used in ICUs globally.

Secondary objectives include assessing the relationship between rehabilitation and key ICU outcomes such as ICU and hospital mortality, length of stay, duration of invasive ventilation, extubation failures, and long-term outcomes including quality of life and functional performance 28 days post-ICU discharge.

The study will also compare rehabilitation practices across different geographic and economic regions to identify potential disparities. The study is structured into three modules, with participation contingent on local resources and feasibility.

The BASIC Module (mandatory for all centers) gathers fundamental data on rehabilitation practices and their association with patient outcomes.

The EXTENDED Module (optional) collects more detailed information on the type, timing, duration, and safety of rehabilitation interventions, including passive exercises, active mobilization, respiratory therapies, dysphagia training, occupational therapy, and cognitive support.

The EXTENDED FOLLOW-UP Module (optional) evaluates the patient's quality of life and functional recovery 28 days after ICU discharge. By examining global rehabilitation practices and their impact on patient outcomes, this study aims to improve rehabilitation strategies in ICUs, contributing to better patient care, recovery, and long-term health outcomes.

DETAILED DESCRIPTION:
* Background --- Critically ill patients often develop intensive care unit (ICU)-acquired weakness (AW), which is defined as clinically detectable weakness without any other plausible explanation. Approximately 40% of these patients experience ICU-AW, associated with higher mortality and long-term morbidity. Early mobilization is an effective rehabilitation strategy that improves both short- and long-term outcomes, reducing hospital stays and enhancing functional recovery. Various rehabilitation interventions-such as mobilization, exercise, respiratory physiotherapy, dysphagia training, occupational therapy, physical activity, and cognitive support-are beneficial but remain underused due to resource limitations. Studies demonstrate improved outcomes with these interventions, emphasizing the role of rehabilitation professionals in the ICU. However, some studies question the effectiveness of these time-consuming and labor-intensive measures, indicating a need for further research. Identifying patient characteristics and detailed intervention information (modality, duration, intensity, frequency) is crucial for effective therapy prescription. The study aims to investigate rehabilitation practices in ICUs globally, focusing on critically ill patients on invasive ventilation who often develop ICU-acquired weakness (ICU-AW). This condition is associated with increased mortality and long-term morbidity. Rehabilitation interventions, including mobilization, physical activity, respiratory physiotherapy, and cognitive support, have shown benefits but remain underutilized.
* Methods --- Study Design and Setting ---- REPOrt is a prospective, international, multicenter, observational cohort study in critically ill invasively ventilated patients, utilizing three modules in which centers can participate, contingent on local capabilities. The practice of rehabilitation can only be studied reliably through a prospective observational study. The study enrollment is planned to start in 2025; the total enrollment period will be 120 days per center. This study will be conducted with the support of the Protective Ventilation Network (PROVE Network) (www.provenetwork.org), in partnership with national and international ICU societies and research institutions. Potentially interested ICUs will be identified. All ICUs that care for adult critically ill invasively ventilated patients can participate in REPOrt. If a hospital has more than one ICU, each ICU can participate as long as patients cared for are adults > 16 years of age (or >18, depending on local rules). The Research Office will handle the list of participating locations as well as the list of primary investigators from each participating institution. Each center interested in participation must submit the study for approval to the local IRB. Adherence to local legislation concerning informed consent will be ensured, including protocols for determining who may provide informed consent in cases where a patient is deemed incapable of doing so themselves. Since this is an observational study, concomitant participation and institutional enrollment in other observation and intervention studies are acceptable.
* Participants --- Patients are eligible for participation if they are admitted to a participating ICU; are adult patients according to local regulations (e.g., aged >16 or >18 depending on local rules); have received invasive ventilation for at least 48 hours; and after written informed consent from the patient or next of kin has been obtained (depending on legislation, and only if rules demand so). Exclusion criteria include withdrawal of life-sustaining treatment.
* Aims of the study and evaluation items --- The primary aim is to describe rehabilitation prevalence and practices in ICUs worldwide. --- Secondary aims include determining the association of rehabilitation and respiratory physiotherapy with typical ICU outcomes, including ICU and hospital length of stay; ICU and hospital mortality; duration of mechanical ventilation, expressed as ventilator-free days and alive at day 28 after ICU admission; and functional outcomes. Additional aims include determining the association of rehabilitation and respiratory physiotherapy with quality of life and functional performance at 28 days after ICU discharge.
* Endpoints --- - Basic information on rehabilitation practices and ICU outcomes (length of stay, duration of ventilation, complications, death). - Granular data on rehabilitative interventions (type, timing, duration, deliverers, safety assessment). - Quality of life and functional performance at 28 days after ICU discharge.
* Data sources and measurements --- Data collected in the study will be captured on an electronic case report form (eCRF) developed in the REDCAP Platform, using an identity code (pseudonym) for patients from countries governed by the General Data Protection Regulation (GDPR) (i.e., European countries). After a patient's eCRF is finalized and approved by the local investigator, anonymization occurs: the identification number is removed, making it impossible to trace back to the patient. Data obtained in the research will be placed immediately into a separate online database for individuals from countries not subjected to the laws.
* Data Collection --- The following data will be collected: - ICU Admission (Day 0): [patient baseline information & pre-hospital status; essential pre-hospital features including SAPS II score; Sequential Organ Failure Assessment (SOFA Score); invasive and non-invasive mechanical ventilation settings; sedation & muscle relaxants; vital signs; temperature; arterial blood gas analysis; delirium and pain assessment; hemodynamic monitoring; general rehabilitation assessment]. - During ICU Stay (Days 0, 3, 7, 14, and ICU discharge): [level of cooperation: S5Q scale; muscle strength using MRC scale; daily intervention duration; types of interventions: passive and active interventions; respiratory physiotherapy specifics; monitoring serious adverse events during interventions]. - ICU Discharge: [outcome assessment: patient pronation; ventilator weaning; airway management; monitoring for any ICU complications]. - 28-Day Follow-Up (Day 28): [post-discharge location; evaluate living arrangements; health assessments; clinical frailty scale; quality of life assessments using the EQ-5D-5L scale; and Modified Rankin Scale (mRS); mortality assessment]. This study is divided into three modules, according to the different aims described above: - BASIC module - to capture basic information on rehabilitation practice worldwide and simple ICU and hospital outcomes, including length of stay in ICU and hospital; duration of ventilation and weaning; airway management; ICU complications, and death. - EXTENDED module - to capture granular data on type, timing, and duration of rehabilitative interventions, who delivers them, and safety assessment. In this module, the focus is on the following rehabilitation interventions: passive interventions (passive exercises, stretching, cycling, electro muscular stimulation, continuous passive motion, etc.); active interventions (exercise therapy, activities of daily living training, mobilization, cycling, etc.); active and passive respiratory physiotherapy (positioning, airways clearance techniques, lung expansion exercises, end-positive airway pressure devices, active cycle of breathing techniques, forced expiratory techniques, assisted or stimulated cough maneuvers, insufflation/exsufflation, inhaled therapy, etc.); and adjunctive techniques (dysphagia training, swallow screening test, cognitive/psychological therapy). - EXTENDED FOLLOW-UP module - to capture quality of life and functional performance at 28 days after ICU discharge.
* Methods for Center Recruitment, Patient Enrollment, and Bias Prevention --- Center Recruitment --- Participating centers will be recruited through a combination of formal private invitations, leveraging established networks from previous studies, and utilizing personal connections within the field of intensive care and rehabilitation. This multi-faceted approach aims to ensure a diverse representation of centers across Europe and beyond, including both large and small institutions.
* Enrollment Strategy --- Invasively ventilated patients will be screened for eligibility over a predefined period of 120 days, with enrollment managed by each center according to local coordinator preferences. Each participating center is expected to enroll between 20 and 40 patients, helping to achieve a comprehensive sample size of approximately 1,200 to 2,400 patients across 60 centers. This range ensures sufficient data to analyze various rehabilitation practices and their clinical outcomes while minimizing the risk of bias.
* Preventing Bias --- To prevent bias from larger centers that may dominate the study, strategies will include: 1) capped enrollment; and 2) diverse center selection.
* Sample Size --- Considering the exploratory nature of this global study and to ensure robust findings, the aim is to enroll approximately 1,200 to 2,400 patients across 60 participating centers. The sample size is based on epidemiological assumption that around 40% of invasively ventilated patients receive rehabilitation. Considering a +/- 2 margin or error, a minimum 2,305 patients are required. Accounting for an anticipated 5% dropout rate, the target enrollment increases to 2,426 patients, which is rounded to 2,400 for practical purposes.
* Statistical Analysis --- A detailed statistical analysis plan is available in the approved protocol.
* Monitoring and Reporting --- National coordinators will oversee the integrity of ethical approval for their country, the data collected, ensuring adherence to standardized protocols and regulations, ensuring compliance with study protocols, and maintaining data integrity. Regular communication will be established among centers to monitor enrollment progress and address any disparities. National coordinators will facilitate communication between centers and provide support for patient enrollment. Each center will designate a lead investigator to oversee local recruitment efforts and ensure accurate data collection. Lead investigators will be responsible for providing ethical approval to the national coordinator and reporting enrollment numbers and any challenges faced during the process.
* Data Validation and Registry Procedures --- To ensure high data quality and reliability of findings, a multi-tiered data validation process will be implemented. These procedures include: 1) Automated data validation rules, including logic checks programmed into the electronic data capture system to validate data entries at the point of data capture: Range checks (e.g., systolic blood pressure between 70-250 mmHg); Format checks (e.g., dates in YYYY-MM-DD format); and Required field enforcement. 2) Manual data review: Periodic manual review of data entries will be conducted by data managers to identify and rectify anomalies not captured by automated rules. 3) Registry access control: Tiered access privileges will be implemented to ensure that only authorized personnel can enter, edit, or approve data.
* Site Monitoring and Auditing --- Site initiation visits may be conducted to train local site teams on study protocols, data entry procedures, and quality expectations if needed. Routine monitoring visits are planned on a remote basis and will occur at regular intervals. Key activities include: 1) Review of source documents; 2) Verification of informed consent processes; 3) Cross-checking data entered into the registry with original records. Audits will be performed to: 1) Verify compliance with study protocol, SOPs, and regulatory requirements; 2) Identify systemic issues and recommend corrective actions
* Data Checks and Consistency Rules --- The data management system will incorporate robust automated checks to identify: 1) Logical inconsistencies (e.g., a male patient marked as pregnant); 2) Temporal inconsistencies (e.g., date of diagnosis after date of death); 3) Missing or duplicate data entries; 4) Interdependent data field checks, ensuring consistency across related variables (e.g., values of Peak pressure on the ventilator above 30 cmH2O or below 10 cmH2O). All detected anomalies will generate queries for site clarification and resolution before data locking in the REDcap system.
* Source Data Verification --- To ensure accuracy and completeness, a proportion of entered data will undergo source data verification, using 1) Random sampling strategy: Some participants will be selected based on enrollment numbers and data risk profiles; 2) Verification process: Comparison of electronic registry (eCRF) data with original case report forms (oCRF), medical records, or other source documentation; 3) Documentation of discrepancies and resolution through a tracked audit trail. Electronic monitoring systems and audit trail logs will be utilized.
* Data Dictionary --- A comprehensive Data Dictionary is available in the appendix of the approved protocol and within each variable in the REDcap system. It will be implemented throughout the study and includes: 1) Variable names and descriptions with clear definitions and purposes of each data element; 2) Coding systems used [e.g., Driving pressure (DP or ΔP) indicates the difference between plateau pressure (Pplat) and positive end-expiratory pressure (PEEP) on the ventilator. Pplat is obtained with an inspiratory pause on the ventilator, to obtain the pressure at the end of inspiration when gas flow has stopped. It is measured in cmH2O]; 3) Acceptable value ranges and units (e.g., mmHg or kPa); 4) Data types and formats. The data dictionary will be updated as needed and made available to all study participants.
* Standard Operating Procedures (SOPs) --- Comprehensive SOPs will guide all aspects of registry operation and ensure consistency and regulatory compliance. Key SOPs include: 1) Patient recruitment and consent: Guidance on ethical and standardized procedures for engaging and enrolling study participants will be guaranteed, with National Coordinators responsible for ensuring consistency and compliance with local regulations; 2) Data collection and entry, including step-by-step instructions for CRF completion with clear definitions, data entry timelines, and handling of missing or ambiguous data; 3) Data management, including data cleaning, validation, backup, and storage; 4) Adverse event reporting, including reportable events, timeframes, and escalation pathways; 5) Monitoring and auditing, including site monitoring schedules, audit plans, and reporting procedures; 6) Change management: amendments to the protocol, CRFs, or registry software, including version control and stakeholder notification will be communicated to all participants regularly.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a participating ICU
* Adult patients (aged 16 years or older, depending on local regulations for the definition of "adults")
* Patients who have received invasive ventilation for at least 48 hours
* Patients who have obtained written informed consent from the patient or next of kin (if local legislation demands so)

Exclusion Criteria:

• Patients admitted for withdrawn of life sustain therapy

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise adult patients admitted to Intensive Care Units (ICUs) located in cities and countries participating in the study.
  Eligible patients will be adult patients requiring invasive mechanical ventilation for at least 48 hours and who can be candidate for rehabilitation during ICU stay.
  Enrolment will be conducted in accordance with applicable local regulations, including the provision of informed consent by the patient or their legally authorized representative.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who received at least one rehabilitation intervention | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Rehabilitation is defined as the delivery of at least one documented intervention during ICU stay, including passive mobilization, active mobilization, or respiratory physiotherapy (active or passive), reported as percentage (%).

SECONDARY OUTCOMES:
Proportion of rehabilitation sessions with at least one Serious Adverse Event (SAE) | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Percentage (%) of rehabilitation sessions with at least one Serious Adverse Event (SAE).
Duration of rehabilitation interventions per day (minutes) | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Duration in minutes of each rehabilitation session, separated into (1) mobilization and (2) respiratory physiotherapy. Minutes per day (median [IQR]).
Proportion of rehabilitation sessions with physiological monitoring | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Monitoring includes electrocardiogram (ECG), peripheral saturation of oxygen (SpO₂), and mean arterial pressure (MAP) measurement during rehabilitation sessions. Binary variables (Yes/No), reported as percentage (%).
Highest level of mobility during ICU stay | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Highest level of mobility measured with the ICU Mobility Scale (IMS). The scale ranges from 0 to 10, with higher scores indicating a higher level of mobility (up to independent walking).
Muscle Strength | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Muscle strength using Medical Research Council (MRC) scale, which evaluates six muscle groups bilaterally (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, ankle dorsiflexion), with each group scored from 0 (no muscle contraction) to 5 (normal strength). The total score ranges from 0 to 60, with lower scores indicating more severe weakness.
ICU length of stay | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Length of stay in the ICU
ICU mortality | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Mortality during ICU stay
ICU complications | From ICU admission (Day 0) until ICU discharge (up to day 28)
  Complications during ICU stay, expressed as percentage (%), defined as neurological complications, infective complications, respiratory complications, deep venous thrombosis, cardiovascular complications, pressure ulcers.
Invasive mechanical ventilation duration during ICU stay | From ICU admission (Day 0) until ICU discharge (up to Day 28)
  Duration of invasive mechanical ventilation during ICU stay
Hospital length of stay | From ICU admission (Day 0) until Hospital discharge (up to Day 365)
  Length of stay in the Hospital
Hospital mortality | From ICU admission (Day 0) until Hospital discharge (up to Day 365)
  Mortality during Hospital stay
Mortality at 28 Days post-ICU discharge | From ICU discharge to Day 28 post-ICU discharge
  Mortality at Day 28
Proportion of patients who received Rehabilitation after ICU discharge at 28 Days post-ICU discharge | From ICU discharge to Day 28 post-ICU discharge
  Any type of rehabilitation (mobilization or respiratory physiotherapy)
Quality of life (EQ-5D-5L scale) at 28 Days post-ICU discharge | From ICU discharge to Day 28 post-ICU discharge
  The Quality of Life outcome will be assessed using EQ-5D-5L scale (Grade 0 to 100) where 0 corresponds to the worst health a patient can immagine and 100 corresponds to best health a patient can immagine.
Clinical Frailty at 28 Days post-ICU discharge | From ICU discharge to Day 28 post-ICU discharge
  The frailty outcome will be assessed using Clinical Frailty Scale (Grade 1 to 9) where 1 corresponds to very fit and 9 corresponds to terminally ill. After ICU discharge until Day 28
Disability at 28 Days post-ICU discharge | From ICU discharge to Day 28 post-ICU discharge
  Disability using modified Rankin Scale (Grade 0 to 6) where 0 indicates no symptoms and 6 indicates patient's death.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Battaglini, MD, PhD, Principal Investigator — Department of Surgical Sciences and Integrated Diagnostics, University of Genoa, Italy; Marcus J Schultz, MD, PhD, Study Chair — Amsterdam University Medical Centers, Amsterdam, The Netherlands; Rik Gosselink, PT, PhD, Study Chair — University of Leuven, Leuven, Belgium; Sabrine N.T. Hemmes, MD, PhD, Study Chair — Amsterdam University Medical Centers, Amsterdam, The Netherlands; Carol L. Hodgson, PhD FACP FAHMS BAppSc(PT) MPhi, Study Chair — Alfred Hospital, Melbourne, VIC, Australia; Ricardo Kenji Nawa, MD, PhD, Study Chair — Hospital Israelita Albert Einstein, São Paulo, SP, Brazil; Irene Schiavetti, PhD, Study Chair — University of Genoa, Italy; Ary Serpa Neto, MD, PhD, Study Chair — Monash University, Melbourne, VIC, Australia; Gentle S. Shrestha, MD, PhD, Study Chair — University Teaching Hospital, Kathmandu, Bagmati, Nepal
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
European regulations for data sharing and privacy

REFERENCES:
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Background] TEAM Study Investigators and the ANZICS Clinical Trials Group; Hodgson CL, Bailey M, Bellomo R, Brickell K, Broadley T, Buhr H, Gabbe BJ, Gould DW, Harrold M, Higgins AM, Hurford S, Iwashyna TJ, Serpa Neto A, Nichol AD, Presneill JJ, Schaller SJ, Sivasuthan J, Tipping CJ, Webb S, Young PJ. Early Active Mobilization during Mechanical Ventilation in the ICU. N Engl J Med. 2022 Nov 10;387(19):1747-1758. doi: 10.1056/NEJMoa2209083. Epub 2022 Oct 26. PMID 36286256
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Van Aerde N, Meersseman P, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Bruyninckx F, Wouters PJ, Gosselink R, Van den Berghe G, Hermans G. Five-year impact of ICU-acquired neuromuscular complications: a prospective, observational study. Intensive Care Med. 2020 Jun;46(6):1184-1193. doi: 10.1007/s00134-020-05927-5. Epub 2020 Jan 22. PMID 31970446
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Appleton RT, Kinsella J, Quasim T. The incidence of intensive care unit-acquired weakness syndromes: A systematic review. J Intensive Care Soc. 2015 May;16(2):126-136. doi: 10.1177/1751143714563016. Epub 2014 Dec 18. PMID 28979394